CLINICAL TRIAL: NCT03074565
Title: Comparison of Ultrasonic Versus Hand Instrumentation Plus Ultrasonic for Effective Sanative Therapy
Brief Title: Ultrasonic Versus Ultrasonic+ for Effective Sanative Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Collaborators: Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery (Other)
Responsible Party: Principal Investigator, Wendy E. Ward, Ph.D., Professor, Brock University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 16-224
Record Dates: First submitted 2017-03-01; First posted 2017-03-09 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Periodontitis; Periodontal Pocket
Keywords: Sanative Therapy; Ultrasonic Therapy; Deep Scaling; Hand Scaling
MeSH Terms: conditions — Periodontitis; Periodontal Pocket | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive one of two treatment modalities on either the left or right side of the mouth on their first treatment visit. During the second treatment visit, subjects will receive the other treatment modality on the other side of the mouth.
Who Masked: Participant, Outcomes Assessor
Masking Description: An investigator, not involved in providing the treatment, will be responsible for randomizing each subject to an initial treatment modality and to which side of the mouth they will receive each treatment. The patient will be masked as to which modality has been used. The care provider cannot be masked as they must use different instrumentation for each treatment type. When assessing outcomes, the investigator will be masked as to the treatment modality and the side of the mouth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonic alone (Experimental): Sanative therapy using ultrasonic instrumentation only.
  Interventions: Device: Ultrasonic alone
- Ultrasonic+ (Active Comparator): Sanative therapy using ultrasonic plus hand instrumentation.
  Interventions: Device: Ultrasonic+

INTERVENTIONS:
Device: Ultrasonic alone — Sanative therapy using ultrasonic instrumentation alone
  Arms: Ultrasonic alone
Device: Ultrasonic+ — Sanative therapy using ultrasonic plus hand instrumentation
  Arms: Ultrasonic+

SUMMARY:
Periodontitis is a chronic oral infection that results in the breakdown of connective tissue and alveolar bone that support the teeth. Non-surgical sanative therapy using a combination treatment of hand and ultrasonic instrumentation is the primary treatment option for patients with periodontitis. However, the hand-held instrumentation requires continuous sharpening for optimal outcomes, which introduces tremendous variability as well as a large increase in time spent by the treating dental hygienists. Therefore, this study aimed to determine if ultrasonic instrumentation alone can provide similar improvements to periodontal outcomes compared to ultrasonic plus hand instrumentation.

DETAILED DESCRIPTION:
Periodontitis is a chronic oral infection that results in the breakdown of connective tissue and alveolar bone that support the teeth. Bacteria and the body's own immune system mediate the severity of periodontitis, where teeth may become loose, fall out or have to be removed. Non-surgical sanative therapy (also referred to as "deep cleaning") is the primary treatment option for patients with generalized chronic periodontitis. This includes debridement with both ultrasonic and hand instrumentation. Using this approach, surgery is avoided for 93% of patients who undergo sanative therapy at our private periodontal specialty practice (unpublished data). However, the hand-held instrumentation requires continuous sharpening for optimal performance, which introduces tremendous variability as well as a large increase in time spent by the hygienists. Ultrasonic instrumentation does not require sharpening, as a new instrument head is used for every new patient.

Therefore, given the interest in "contemporary instrumentation", meaning ultrasonic therapy alone, the primary objective of this study is to determine if similar improvements in periodontal indices can be achieved using ultrasonic instrumentation alone versus ultrasonic instrumentation in conjunction with hand instrumentation.

Secondary objectives included the following: i) to determine if the time required to complete sanative therapy is reduced using ultrasonic therapy alone, given the ultrasonic instruments do not require sharpening and less instrument changes by the hygienist are required during treatment. If the time is less for ultrasonic therapy alone, there is a potential cost-savings for the patient, as well as less time spent receiving therapy in the dental chair; ii) to determine if the treatment with ultrasonic therapy versus ultrasonic therapy and hand instrumentation is more comfortable for the patient; and iii) to determine if there is less sensitivity to the teeth with ultrasonic therapy alone compared to the combination of ultrasonic therapy and hand instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females age 19 years or older who are undergoing sanative therapy for moderate to severe chronic periodontitis are eligible.
* Chronic periodontitis has been classified as localized or generalized depending on whether <30% or >30% of sites are involved.
* Severity is based on the amount of clinical attachment loss (CAL) and is designated as slight (1-2 mm CAL), moderate (3-4 mm CAL) or severe (> 5 mm CAL).

Exclusion Criteria:

* Patients with dental implants,
* pregnancy,
* a recent history of antibiotic use (within 3 months prior to treatment) and
* inability to give consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Periodontal healing evaluated based on changes in mean probing depth (mm) | Baseline and between 8 and 12 weeks after sanative therapy
  Healing is evaluated based on changes in mean probing depth

SECONDARY OUTCOMES:
Plaque index | Baseline and between 8 and 12 weeks after sanative therapy
  O'Leary Plaque Score Index is a score in the total amount of plaque present at 4 surfaces of a tooth
Bleeding on Probing | Baseline and between 8 and 12 weeks after sanative therapy
  Inflammation is determined by percent of bleeding sites that are measured at 6 sites per tooth
Clinical Attachment Loss (Periodontal Attachment Loss) | Baseline and between 8 and 12 weeks after sanative therapy
  Periodontal healing is evaluated based on changes in clinical attachment loss

OTHER OUTCOMES:
Time spent | Average sanative therapy session is 90 minutes
  Time spent receiving treatment with either modality
Comfort of the experience | Average sanative therapy session is 90 minutes
  The level of comfort experienced by the patient during treatment
Tooth sensitivity | Sanative therapy appointment (90 minutes) and 8 to 12 weeks after sanative therapy
  The level of tooth sensitivity experienced by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Fritz, D.D.S., Study Director — Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery
Locations (2):
- Canada (2):
  - Dr. Peter C. Fritz, Reconstructive Periodontics and Implant Surgery, Fonthill, Ontario
  - Brock University, St. Catharines, Ontario

IPD SHARING:
Plan to Share IPD: No